CLINICAL TRIAL: NCT01245634
Title: Study Assessing 20 mg/kg Dose of the Recombinant Human Monoclonal Antibody Against P-selectin in Patients Undergoing Coronary Artery Bypass Graft (CABG) Surgery
Brief Title: A Study of RO4905417 in Patients Undergoing Coronary Artery Bypass Graft (CABG) Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BP25601
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Coronary Heart Disease, Graft Occlusion, Vascular
MeSH Terms: conditions — Coronary Disease | interventions — inclacumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental)
  Interventions: Drug: RO4905417
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — iv infusion every 4 weeks, 32 weeks
  Arms: B
Drug: RO4905417 — 20 mg/kg iv infusion every 4 weeks, 32 weeks
  Arms: A

SUMMARY:
This randomized double-blind, placebo-controlled study will evaluate the efficacy and safety of RO4905417 in the prevention of saphenous vein graft disease in patients undergoing elective or urgent coronary artery bypass (CABG) surgery. Patients will be randomized to receive either RO4905417 20 mg/kg by intravenous infusion or placebo every 4 weeks for 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, > 18 and > 85 years of age
* Patients undergoing primary multi-vessel CABG with at least one saphenous vein graft. with or without cardiopulmonary bypass
* Body mass index (BMI) </= 35 kg/m2

Exclusion Criteria:

* Participation in previous studies evaluating RO4905417
* Positive for HIV, receiving antiretroviral drugs, or immuno-suppressed
* Acute infection at screening or active chronic infection within 3 months prior to CABG surgery
* Patients undergoing emergency cardiac surgery for an immediately life-threatening condition
* Patients undergoing concomitant valve surgery
* History of CABG (only patients without prior CABG surgery will be admitted to the study)
* Left ventricular ejection fraction < 20%
* History of transient ischemic attack or stroke within the 12 weeks prior to the CABG procedure
* Significant renal or liver impairment
* Malignancy diagnosed within the previous 5 years (except for successfully resected basal cell cancer)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2010-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with diameter stenosis >50% (including total occlusion) of at least one saphenous vein graft, as assessed by invasive angiography | 1 year

SECONDARY OUTCOMES:
Lumen diameter of saphenous vein grafts, as assessed by invasive angiography | 1 year
Proportion of patients needing revascularization | 1 year
Safety: Incidence of adverse events (including major adverse cardiovascular events) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (30):
- United States (24):
  - Huntsville, Alabama
  - Tucson, Arizona
  - Los Angeles, California
  - Atlantis, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Macon, Georgia
  - Springfield, Illinois
  - Fort Wayne, Indiana
  - Lexington, Kentucky
  - Dearborn, Michigan
  - Petoskey, Michigan
  - Royal Oak, Michigan
  - Troy, Michigan
  - Duluth, Minnesota
  - Saint Paul, Minnesota
  - Washington, Missouri
  - Stony Brook, New York
  - Durham, North Carolina
  - Toledo, Ohio
  - Memphis, Tennessee
  - Dallas, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
- Canada (6):
  - Saint John, New Brunswick
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec

REFERENCES:
- [Derived] Stahli BE, Tardif JC, Carrier M, Gallo R, Emery RW, Robb S, Cournoyer D, Blondeau L, Johnson D, Mann J, Lesperance J, Guertin MC, L'Allier PL. Effects of P-Selectin Antagonist Inclacumab in Patients Undergoing Coronary Artery Bypass Graft Surgery: SELECT-CABG Trial. J Am Coll Cardiol. 2016 Jan 26;67(3):344-6. doi: 10.1016/j.jacc.2015.10.071. No abstract available. PMID 26796402